CLINICAL TRIAL: NCT06729762
Title: Ultrasound-guided Thermal Ablation for the Treatment of Benign Thyroid Nodules: A Multicenter Study
Brief Title: Ultrasound-guided Thermal Ablation for Benign Thyroid Nodules
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu-kun Luo, Clinical Professor, Chinese PLA General Hospital
Other Study IDs: 2024-654
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Nodule (Benign)
MeSH Terms: conditions — Thyroid Nodule | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- ultrasound-guided thermal ablation: ultrasound-guided thermal ablation
  Interventions: Procedure: ultrasound-guided thermal ablation

INTERVENTIONS:
Procedure: ultrasound-guided thermal ablation — radiofrequency ablation, microwave ablation, laser ablation

SUMMARY:
To evaluate long-term outcomes of ultrasound-guided thermal ablation for benign thyroid nodules

DETAILED DESCRIPTION:
To evaluate and predict long-term clinical outcomes of ultrasound-guided thermal ablation for benign thyroid nodules by a multicenter study

ELIGIBILITY:
Inclusion Criteria:

1. confirmation of benign nodule status on two separate fine- needle aspiration or core-needle biopsy
2. no suspicious malignant features on ultrasound examination
3. report of cosmetic and/ or symptomatic problems or concern of nodules growing rapidly or malignant transformation
4. refusal or ineligibility for surgery
5. follow-up time ≥12 months

Exclusion Criteria:

1. follicular neoplasm or malignancy findings on biopsy
2. nodules with benign result on biopsy had suspicious of malignancy in US
3. patients with contra-lateral vocal cord paralysis
4. previous radiation to the head and neck
5. follow- up time less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with thyroid nodules
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
volume reduction rate | through study completion, an average of 6 months
  The volume reduction rate (VRR)was calculated by the equations: VRR=([initial volume-final volume] × 100)/initial volume

SECONDARY OUTCOMES:
rate of complications | 1 week
  complications after ablation
cosmetic score | through study completion, an average of 6 months
  The cosmetic score was assessed by a physician (1, no palpable mass; 2, no cosmetic problem but palpable mass; 3, a cosmetic problem on swallowing only; and 4, a readily detected cosmetic problem)
symptom score | through study completion, an average of 6 months
  The symptom score was self-measured by patients using a 10-cm visual analogue scale (grade 0-10)
rate of nodule regrowth | through study completion, an average of 6 months
  Regrowth was defined as ≥50% volume increase compared to the previously recorded smallest volume during the follow-up
rate of change of thyroid function | through study completion, an average of 6 months
  thyroid function test, including free triiodothyronine, free thyroxine, thyroid stimulating hormone, thyroid peroxidase antibody and anti-thyroglobulin antibodies
rate of disappearance | through study completion, an average of 6 months
  complete disappearance of ablated nodule on ultrasound and contrast-enhanced ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Yukun Luo, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No